CLINICAL TRIAL: NCT02700685
Title: Effect of a Polyphenol-rich Plant Extract on Attention-Deficit Hyperactivity Disorder (ADHD): A Randomized, Double Blind, Placebo and Active Product Controlled Multicenter Trial.
Brief Title: Effect of Pycnogenol® on ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nina Hermans (Other)
Responsible Party: Sponsor-Investigator, Nina Hermans, Prof. Dr., Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pycno 2015-14
Record Dates: First submitted 2016-01-18; First posted 2016-03-07 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pycnogenols; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pycnogenol (Experimental): Dietary supplement, standardised extract of French maritime Pine bark. This group receives a nutritional supplement for a period of 10 weeks.
  Subjects < 30 kg body weight: 20 mg Pycnogenol/day Subjects >= 30 kg body weight: 40 mg Pycnogenol/day
  Interventions: Dietary Supplement: Pycnogenol
- Placebo (Placebo Comparator): Placebo treatment (identical capsules containing excipients only)
  Interventions: Other: Placebo
- Methylphenidate (Active Comparator): Standard pharmaceutical treatment for ADHD, slow release. Subjects < 30 kg body weight: 20 mg methylphenidate once per day Subjects >= 30 kg body weight: 30 mg methylphenidate once per day
  Interventions: Drug: Methylphenidate

INTERVENTIONS:
Dietary Supplement: Pycnogenol — Dietary supplement, standardised extract of French maritime Pine bark. This group receives a nutritional supplement for a period of 10 weeks.
  Arms: Pycnogenol
Drug: Methylphenidate — Standard pharmaceutical treatment for ADHD, slow release.
  Arms: Methylphenidate
Other: Placebo — Placebo treatment (identical capsules containing excipients only)
  Arms: Placebo

SUMMARY:
This double blind, randomised controlled trial examines the effect of a commercially available nutritional supplement on behaviour of ADHD patients, as well as on their physical and psychiatric co-morbidities, and level of oxidative stress and immune activity, as compared to placebo and standard pharmaceutical treatment for ADHD.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 6-12 years old (both inclusive).
* The patient satisfies the DSM-IV criteria for ADHD or ADD.
* The patient has a responsible caregiver who is able to provide information about the patient's functional status.
* Written informed consent is obtained from the patient and the legally accepted representative.

Exclusion Criteria:

* The patient does satisfy the DSM-IV for autism spectrum disorder.
* The patient does have situational hyperactivity, pervasive developmental disorders, schizophrenia, other psychotic disorders such as mood or anxiety disorder, personality disorder as unsocial behaviour, personality change due to a general medical condition, mental retardation (IQ < 70), understimulating environments, conduct disorder, chorea and other dyskinesias. The patient does not have tics or Tourette's syndrome, or personal or family history of psychotic disorder, bipolar illness, depression, or suicide attempt.
* The patient does have any chronic medical disorder (diabetes, epilepsy or other seizure disorder, autoimmune disorder, gastrointestinal disorder, renal or cardiovascular disorders, etc.) or acute inflammatory disease. The patient does not have glaucoma, heart disease, heart rhythm disorder, high blood pressure, or peripheral vascular disease such as Raynaud's syndrome.
* The patient did use any of these medications during the 3 months before entering the study: clonidine, guanethidine, blood thinners (e.g. warfarin or Coumadin), antidepressants (e.g. amitriptyline, citalopram, doxepin, fluoxetine, nortriptyline, paroxetine, sertraline), cold or allergy medicine that contains a decongestant, medications to treat high or low blood pressure, seizure medicine (e.g. phenobarbital, phenytoin, primidone), or diet pills.
* The patient did take MAO inhibitor (isocarboxazid, linezolid, phenelzine, rasagiline, selegiline or tranylcypromine) in the past 14 days.
* The patient has any other contraindication for the use of methylphenidate.
* The patient did use vitamin/mineral/herbal/omega-3 supplements or other any medication (psychoactive medication, antibiotics, anti-inflammatory drugs, melatonin, etc.) > 1 week during the 3 months before inclusion.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Summed ADHD score of the ADHD-Rating Scale as rated by teachers | 10 weeks

SECONDARY OUTCOMES:
Summed ADHD score of the ADHD-Rating Scale as rated by teachers | 5 weeks
Summed ADHD score of the ADHD-Rating Scale as rated by parents | 5 weeks, 10 weeks
Summed ADHD score of the Social-Emotional Questionnaire (SEQ) as rated by parents and teachers | 10 weeks
Scores on ADHD subscales of the ADHD-RS as rated by parents and teachers - hyperactivity, impulsivity and inattention | 5 & 10 weeks
Scores on ADHD subscales of the SEQ as rated by parents and teachers - hyperactivity, impulsivity and inattention | 5 & 10 weeks
Percentage of responders (ADHD-RS) as rated by parents and teachers | 5 & 10 weeks
  Score reduction of at least 20% for parents and/or teachers
Percentage of responders (SEQ) as rated by parents and teachers | 5 & 10 weeks
  Score reduction of at least 20% for parents and/or teachers
Social behavior problems subscale of the SEQ, as rated by parents and teachers | 10 weeks
Anxiety subscale of the SEQ, as rated by parents and teachers | 10 weeks
Physical and sleep complaints score as measured by the Physical Complaints Questionnaire (PCQ) | 5 & 10 weeks
Erythrocyte glutathione (GSH) level | 10 weeks
Urinary 8-OHdG level | 10 weeks
Plasma cytokine levels | 10 weeks
Plasma antibody levels | 10 weeks
Gene expression | 10 weeks
Serum neuropeptide Y | 10 weeks
Serum zinc | 10 weeks
Intestinal microbial composition | 10 weeks
Intervention acceptability | 10 weeks
  Percentage of participants with side effects, treatment adherence and proportion of drop-outs
Intervention acceptability | 10 weeks
  Percentage of participants with side effects
Intervention acceptability | 10 weeks
  Proportion of drop-outs
Intervention acceptability | 10 weeks
  Treatment adherence
Urinary catecholamines | 10 weeks
Plasma lipid-soluble vitamins | 10 weeks
Long-term follow up | 6 months
  Long-term follow up on eventual treatment choice (medication, no intervention, nutritional supplement)
Long-term follow up | 6 months
  Long-term follow up on behaviour
Long-term follow up | 6 months
  Long-term follow up on physical/psychiatric complaints

CONTACTS AND LOCATIONS:
Overall Officials: Nina Hermans, PhD, Study Director — Universiteit Antwerpen
Locations (3):
- Belgium (3):
  - Universitaire Kinder- en Jeugdpsychiatrie, Borgerhout
  - University Hospital Antwerp, Edegem
  - University Hospital Ghent, Ghent

REFERENCES:
- [Derived] Verlaet AA, Ceulemans B, Verhelst H, Van West D, De Bruyne T, Pieters L, Savelkoul HF, Hermans N. Effect of Pycnogenol(R) on attention-deficit hyperactivity disorder (ADHD): study protocol for a randomised controlled trial. Trials. 2017 Mar 28;18(1):145. doi: 10.1186/s13063-017-1879-6. PMID 28351412